CLINICAL TRIAL: NCT00251056
Title: A Phase IIa Randomised, Open Label, Dose Response Study to Determine the Optimum Dose of Dry Powder Mannitol Required to Generate Clinical Improvement In Patients With Cystic Fibrosis
Brief Title: Mannitol Dose Response Study in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Brett Charlton, Pharmaxis Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DPM-CF-202
Record Dates: First submitted 2005-06-30; First posted 2005-11-09 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: mannitol
- 2 (Active Comparator)
  Interventions: Drug: mannitol
- 3 (Active Comparator)
  Interventions: Drug: mannitol
- 4 (Active Comparator)
  Interventions: Drug: mannitol

INTERVENTIONS:
Drug: mannitol — 120mg BD
  Arms: 2
Drug: mannitol — 40 mg BD
  Arms: 1
Drug: mannitol — 240mg BD
  Arms: 3
Drug: mannitol — 400mg BD
  Arms: 4

SUMMARY:
Many cystic fibrosis patients die of lung failure caused by repeated lung infections from thick, sticky mucus. Past studies have shown Bronchitol inhalation may help to facilitate the clearance of mucus by altering its rheology and replenishing the airway surface liquid layer in these patients, thereby enhancing the shift of stagnant mucus from the lungs. The study aim is to determine the optimal dose of mannitol to generate clinical improvement in patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis (sweat test/genotype)
* 7 years or older
* FEV1 between 40% and 90% of predicted for height, age and gender.
* Able to perform acceptable-quality spirometry
* Clinically stable in the week up to study entry
* No additional antibiotics or additional oral steroids for a period of 14 days before study entry (routine antibiotics permitted)

Exclusion Criteria

* Currently active asthma
* Subjects colonized with Burkholderia cepacia or MRSA
* Considered "terminally ill" or listed for transplantation
* Requiring home oxygen or assisted ventilation
* Concurrent illness that in the investigators opinion may contribute to an increased and unacceptable risk if the subject was enrolled in the study (e.g. significant varicies, portal hypertension, cor pulmonale)
* Significant episode of haemoptysis (>60 mLs) in the previous 12 months
* Heart attack or stroke in last 3 months
* Known aortic or cerebral aneurysm
* Subjects who are breast feeding or pregnant.
* At risk females unwilling to use appropriate contraception to prevent pregnancy during the course of the study
* Subjects who have participated in another investigative drug study parallel to, or within 4 weeks of study entry.
* Known intolerance to mannitol or unable to take any form of bronchodilator medications.
* Uncontrolled hypertension, systolic BP > 200 or diastolic BP> than 100
* Concurrent use of beta blocker medication
* Concurrent use of hypertonic saline

Canada:

* Concurrent use of other pharmacological mucolytic agents other than Pulmozyme

Argentina:

* Concurrent use of other pharmacological mucolytic agents including Pulmozyme

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
FEV1 | 2 weeks
FVC | 2 weeks

SECONDARY OUTCOMES:
other measures of lung function | various
QOL | 2 weeks
sputum microbiology | 2 weeks
safety | 2 weeks
sputum clearance and cough | 2 weeks
respiratory symptoms | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Tullis, MD, Principal Investigator — St Michaels Hospital, Toronto, Ontario, Canada; Brett Charlton, MBBS PhD, Study Director — Pharmaxis Ltd, Sydney, NSW, Australia
Locations (12):
- Argentina (5):
  - Hospital de Niños Superiora Sor María Ludovica, La Plata, Buenos Aires
  - Hospital Pediatrico, Resistencia, Chaco Province
  - Hospital Interzonal Especializado Materno Infantil (HIEMI), Buenos Aires
  - Hospital General de Niños, CABA
  - Hospital Pediatrico Dr Humberto J Notti, Mendoza
- Canada (7):
  - BC Children's Hospital, Vancouver, British Columbia
  - St Pauls Hospital, Vancouver, British Columbia
  - Janeway Children's Health and Rehabilitation Center, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - St Michaels Hospital, Toronto, Ontario